CLINICAL TRIAL: NCT00001414
Title: Mapping Personality Traits to Genes
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 940122; 94-M-0122
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-06

CONDITIONS: Mental Disorder
Keywords: Behavior Genetics; Normal Personality; Intelligence; Siblings; Sixteen Personality Factor Questionnaire; NEO-Personality Inventory (Revised); X-Chromosome
MeSH Terms: conditions — Mental Disorders

SUMMARY:
Previous research involving families, twins, and adoption all support the idea that there is a substantial heritable aspect to personality.

The goal of this research study is to determine how genetics influence heritable personality traits. The work will focus on how genetics affect the chemical messengers which brain cells use to communicate with each other (neurotransmitters).

The study involves collecting personality data and DNA samples from related individuals, primarily male siblings and female siblings, but also including parents. Genetic tests performed on these samples will continue to focus on variations in genes, which potentially effect brain neurotransmission.

This research has the potential to advance knowledge of genetic influences on human behavior that may be relevant both to normal personality and to psychopathology.

DETAILED DESCRIPTION:
Building on family, twin and adoption studies suggesting that substantial aspects of personality are heritable, research under this protocol explores potential genetic influences on normal personality dimensions. We have previously reported associations between variation in neurotransmitter system genes and variation in personality traits, both across and within families, in a sample of the general population. This study involves collecting personality data and DNA samples from related individuals, primarily male siblings and female siblings, but also including parents. Genetic tests performed on these samples will continue to focus on variations in genes, which potentially affect brain neurotransmission. In some cases, participants are recontacted to specifically investigate whether identified variations in neurotransmitter system genes actually affect neurotransmission. Large population samples are needed in this research, particularly since a new epidemiologically standard population sample will be obtained. This research has the potential to advance knowledge of genetic influences on human behavior that may be relevant both to normal personality and to psychopathology.

ELIGIBILITY:
Personality data and DNA samples will be collected from related individuals, primarily pairs of male and pairs of female siblings, but also including parents.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2400
Dates: Start 1994-04; Study Completion 2002-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Ahern FM, Johnson RC, Wilson JR, McClearn GE, Vandenberg SG. Family resemblances in personality. Behav Genet. 1982 May;12(3):261-80. doi: 10.1007/BF01067847. No abstract available. PMID 6889860
- [Background] Amos CI, Elston RC, Wilson AF, Bailey-Wilson JE. A more powerful robust sib-pair test of linkage for quantitative traits. Genet Epidemiol. 1989;6(3):435-49. doi: 10.1002/gepi.1370060306. PMID 2753353
- [Background] Benjamin J, Li L, Patterson C, Greenberg BD, Murphy DL, Hamer DH. Population and familial association between the D4 dopamine receptor gene and measures of Novelty Seeking. Nat Genet. 1996 Jan;12(1):81-4. doi: 10.1038/ng0196-81. No abstract available. PMID 8528258